CLINICAL TRIAL: NCT02732704
Title: THE ALIGN-AR TRIAL: Safety and Effectiveness/Performance of the Transfemoral JenaValve Pericardial TAVR System in the Treatment of Patients With Symptomatic Severe Aortic Regurgitation (AR)
Brief Title: THE ALIGN-AR EFS TRIAL: JenaValve Pericardial TAVR Aortic Regurgitation Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JenaValve Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0004; P02C320_JV06EFS_CIP (Other: JenaValve Technology Inc.); CA-0002 EU (Other: JenaValve Technology Inc.); CA-0002 Germany (Other: JenaValve Technology Inc.); CA-0011 (Other: JenaValve Technology Inc.)
Record Dates: First submitted 2016-03-18; First posted 2016-04-11 (Estimated); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Aortic Regurgitation
Keywords: Aortic Valve Disease; Aortic Regurgitation; Aortic Insufficiency
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transcatheter Aortic Valve Replacement (TAVR) (Experimental): TAVR with JenaValve Pericardial Valve and Delivery System
  Interventions: Device: JenaValve Pericardial TAVR System

INTERVENTIONS:
Device: JenaValve Pericardial TAVR System — TAVR with JenaValve Pericardial Valve and Delivery System

SUMMARY:
To collect information about treatment for severe Aortic Regurgitation (AR), which affects the aortic valve in the heart. Aortic regurgitation is a condition where aortic valve in the heart does not close tightly and allows some blood to leak back into the heart chamber. Symptoms of aortic regurgitation may include fatigue and shortness of breath. The preferred treatment for severe aortic regurgitation is aortic valve replacement surgery.

DETAILED DESCRIPTION:
This study will examine the use of TAVR (Transcatheter Aortic Valve Replacement), which is a minimally invasive procedure designed to replace the aortic valve inside the heart. In this study, TAVR will be performed using the JenaValve Pericardial TAVR System, which is intended to help treat severe aortic regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with severe aortic regurgitation (AR).
* Patient at high risk for open surgical valve replacement
* Patient symptomatic according to NYHA functional class II or higher
* The study patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB)/ Ethics Committee (EC) of the respective clinical site.

Exclusion Criteria:

* Congenital uni or bicuspid aortic valve morphology
* Previous prosthetic aortic valve (bioprosthesis or mechanical) implant
* Endocarditis or other active infection
* Need for urgent or emergent TAVR procedure for any reason
* Cardiogenic shock or hemodynamic instability requiring inotropic support or ventricular assist device
* Severe mitral regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-20 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality at 30 days | 30 days
  All-Cause mortality within the first 30 days post index procedure

SECONDARY OUTCOMES:
Mortality | At 30 days
  Absence of procedural mortality
Peri-Procedural Myocardial Infarction | At ≤72hr after the index procedure
  Peri-procedural and spontaneous myocardial infarction
Stroke-Free Survival | At 30 days and 1 year
  Disabling or non-disabling stroke
Bleeding & Vascular Complications | 30 days
  Major and minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Martin B. Leon, MD, Study Chair — New York-Presbyterian/ Columbia University Medical Center; Torsten P. Vahl, MD, Principal Investigator — New York-Presbyterian/ Columbia University Medical Center; Vinod H. Thourani, MD, Principal Investigator — Piedmont Healthcare; Stephan Baldus, MD, Principal Investigator — Herzzentrum der Universität zu Köln
Locations (19):
- United States (9):
  - Cedars Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Piedmont Healthcare, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - New York-Presbyterian/ Columbia University Medical Center, New York, New York
  - Baylor Scott & White Research Institute, Dallas, Texas
  - University of Washington, Seattle, Washington
- Germany (7):
  - Kerckhoff-Klinik GmbH Bad Nauheim, Bad Nauheim
  - Herz- und Diabeteszentrum NRW Ruhr-Universität Bochum Bad Oeynhausen, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Herzzentrum der Universität zu Köln, Cologne
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitäres Herzzentrum Hamburg, Hamburg
- Netherlands (3):
  - Leiden University Medical Center, Leiden
  - St. Antonius Hospital, Nieuwegein
  - Erasmus University Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamid N, Ranard LS, Khalique OK, Hahn RT, Nazif TM, George I, Ng V, Leon MB, Kodali SK, Vahl TP. Commissural Alignment After Transfemoral Transcatheter Aortic Valve Replacement With the JenaValve Trilogy System. JACC Cardiovasc Interv. 2021 Sep 27;14(18):2079-2081. doi: 10.1016/j.jcin.2021.07.025. No abstract available. PMID 34556282